CLINICAL TRIAL: NCT05174260
Title: Predictability of Hemodynamic Instability With Increase in Perfusion Index (PI) and Pleth Variability Index (PVI) Values After Spinal Block in Elective Cesarean Sections
Brief Title: The Relationship Between Perfusion Index and Pleth Variability Index and Hemodynamics in Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, ESMA KAPLAN ÇALIŞKAN, assistant doctor, Adiyaman University
Other Study IDs: date:18/05/2021 ID:2021/05-23; öznur uludağ (Other: Adıyaman university)
Record Dates: First submitted 2021-11-08; First posted 2021-12-30 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Effects of Anesthesia Spinal and Epidural in Pregnancy
Keywords: spinal anesthesia; perfusion index
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypotension developing group: Pregnant women who underwent elective C/S under spinal anesthesia with systolic arterial pressure below 90 mmHg or with hypotension symptoms such as dizziness, nausea and vomiting during the procedure.
  Interventions: Device: perfusion index, pleth variable index
- group without hypotension: Pregnant women who underwent elective cesarean section under spinal anesthesia whose systolic arterial pressure did not fall below 90 mmHg or did not have any symptoms of hypotension during the procedure.
  Interventions: Device: perfusion index, pleth variable index

INTERVENTIONS:
Device: perfusion index, pleth variable index — a clip will be attached to the patient's finger and the perfusion index and pvi will be measured
  Other Names: a latch will be attached to the patient's finger

SUMMARY:
In routine practice, the preferred anesthesia method in cesarean section operations is spinal anesthesia, but it causes hypotension in a significant part of the patients. In this study, the researchers planned to evaluate the perfusion index (PI) and pleth variability index (PVI) values at different positions to predict hypotension after spinal anesthesia applied for cesarean section. When hypotension is severe and persistent, it may cause uteroplacental perfusion disorder, fetal hypoxia-acidosis, and neonatal neurological damage as well as nausea-vomiting, loss of consciousness, cardiac arrest and collapse in the mother(2) If hemodynamic changes such as hypotension and bradycardia are present, symptoms may occur. . Early intervention with vasoconstrictor agents will be provided to prevent the emergence of the disease, disturbing symptoms and other complications that may occur will be prevented.

DETAILED DESCRIPTION:
In recent years, the trend towards noninvasive monitoring methods has increased instead of invasive monitoring methods. Plet Variability Index (PVI), perfusion index (PI) are non-invasive, easily applicable and easily interpretable new monitoring methods. It has been shown that intraoperative hypotension and fluid requirement can be predicted, especially with Plet Variability Index (PVI) monitoring. Hypotension is the most common complication of spinal anesthesia. If no precautions are taken, it is seen in 80-90% of cases. associated with a decrease in peripheral vascular resistance. Recent studies have shown that cardiac output does not decrease, but slightly increases or does not change, and venous return does not change with spinal anesthesia. Aortocaval compression may exacerbate hypotension due to neuraxial anesthesia. The PI is obtained by calculating the ratio of pulsatile blood flow to nonpulsatile blood flow in peripheral tissues by pulse oximetry. This ratio reflects changes in peripheral vascular resistance. For example, a low PI indicates peripheral vasoconstriction. PVI represents changes in PI that occur during one or more complete respiratory cycles. Provides evaluation of intravascular volume; and a higher PVI is associated with greater responsiveness to fluid volumes. In some studies, it is stated that PI and PVI values obtained from pulse oximetry are predictive for SA-induced hypotension in cesarean deliveries; There are also studies in the literature showing the opposite. In this study, the researchers aimed to test the hypothesis that hypotension can be predicted by using PVI representing cardiac preload and PI representing vascular tone in pregnant women after spinal anesthesia and to examine the superiority of these values.

OBJECTIVE: Today, spinal anesthesia (SA); Since it is less risky for maternal and new born health compared to general anesthesia, it is a more preferred method in elective cesareansection operations. Hypotension due to spinal anesthesia, which is the most common side effect of spinal anesthesia, is frequently seen in patients. Due to the negative consequences of hypotension on the mother and newborn; It is important to take the necessary precautions against this hemodynamic deterioration. Perfusion index (PI) and pleth variability index (PVI) are parameters that can be measured noninvasively by pulseoximetry. In our study; By examining the lower extremity PI and PVI values in patients who will undergo elective cesareansection with SA; We investigated the usability and superiority of these values over each other in predicting hemodynamic deterioration.

METHODS: This research; It was conducted as a prospective observational study and 113 pregnant women aged 18-40 years who were ASA1-2 who were going to undergo lower segment cesarean section were included in our study. Demographic data of the patients (age, gender, weight, height, BMI) and routine hemogram values (hemoglobin, hematocrit, platelet, wbc) taken for preoperative evaluation were recorded. After the patients were placed on the operating table, PI and PVI values in the supine and sitting positions, PI and PVI values at the 1st, 2nd, 3rd, and 4th minutes after spinal anesthesia was applied to the patient, and finally, the postpartum PI, PVI values were recorded. In addition, in order to follow up the hemodynamic changes in all patients in thes tudy, Standard monitoring including electrocardiography, non-invasive blood pressure measurements and pulse measurement was performed, and changes in systolic pressure, diastolic pressure and heart rate were recorded before and after spinal anesthesia.

In our study, in which we examined PI and PVI values in predicting hypotension due to spinal anesthesia in elective C/S operations, we have reached the following results.

Unlike other studies in the literature; In our study, in which we followed the PI and PVI values in the lower extremities together and examined the diagnostic superiority of these values to each other and the relationship between the hemogram and hematocrit values of the patients, we did not find a statistically significant difference in the increase in the lower extremity basal PI and PVI values in the patient groups with and without hypotension. We interpreted this situation as lower extremity basal PI and PVI values were not effective in predicting hypotension due to spinal anesthesia.

We observed that there was no change in PI and PVI values in 5 patients who were not included in the study in whom spinal anesthesia failed, and that there was an increase in successful procedures independent of the development of significant hemodynamic instability. As a result, our study supported previous studies that PI and PVI values could be used to evaluate the success of spinal block.

In addition, we found that hgb and hct values were significantly lower in the hypotension-developing group in our study, but we found that this did not cause a significant difference in basal PI and PVI values. We think that the surgical HGB limit should be reconsidered in patients who will undergo elective surgery, due to the increased risk of hypotension if the patients have low hemogram values, and we believe that it would be beneficial to conduct more comprehensive multicenter studies in both cases.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who will undergo elective cesarean section
2. Patients with ASA 1-2
3. Patients aged 18-40 years

Exclusion Criteria:

1. Emergency cases
2. <18 or > 40 years old
3. Gestational age <36 weeks
4. BMI ≥40
5. Cardiovascular disease
6. Patients with ASA 3-4
7. Those with peripheral vascular disease
8. Patients for whom spinal anesthesia is contraindicated
9. Refusal to participate

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients aged 18-40 who will undergo elective cesarean section
Sampling Method: Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
perfusion index (PI) | perioperative
  Before and after spinal anesthesia, 4 measurements will be made until the baby is born, and 1 more measurement will be made after routine oxytocin. Its relationship with hemodynamic deterioration will be examined and compared between both groups.In basal values of PI and the rate of change of these values; There was no significant difference between the groups with and without hypotension.
pleth variability index (PVI) | perioperative
  Before and after spinal anesthesia, 4 measurements will be made until the baby is born, and 1 more measurement will be made after routine oxytocin. Its relationship with hemodynamic deterioration will be examined and compared between both groups.In basal values of PVI and the rate of change of these values; There was no significant difference between the groups with and without hypotension.
BMİ-weight, | preoperratif value
  There was no difference in BMI and weight values between patients who developed and did not develop hypotension after spinal anesthesia
hemoglobin | preoperatif value
  Hemoglobin (p=0.014) and hematocrit (p=0.012) values weres ignificantly lower in pregnant women who developed hypotension
APGAR | the 1st minute APGAR-the 5th minute APGAR
  The 1st minute APGAR (p=0.005= and 5th minute APGAR (p=0.014) scores were significantly lower in the babies of pregnant women who developed hypotension.

SECONDARY OUTCOMES:
systolic blood pressure | perioperative
  systolic blood pressure will be recorded
diastolic blood pressure | perioperative
  diastolic blood pressure will be recorded
pulse | perioperative
  pulse will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I am undecided about sharing individual participant data with other researchers.

REFERENCES:
- [Background] Loubert C. Fluid and vasopressor management for Cesarean delivery under spinal anesthesia: continuing professional development. Can J Anaesth. 2012 Jun;59(6):604-19. doi: 10.1007/s12630-012-9705-9. Epub 2012 Apr 24. English, French. PMID 22528166
- [Background] Langesaeter E, Rosseland LA, Stubhaug A. Continuous invasive blood pressure and cardiac output monitoring during cesarean delivery: a randomized, double-blind comparison of low-dose versus high-dose spinal anesthesia with intravenous phenylephrine or placebo infusion. Anesthesiology. 2008 Nov;109(5):856-63. doi: 10.1097/ALN.0b013e31818a401f. PMID 18946298
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Result] Tsuchiya M, Yamada T, Asada A. Pleth variability index predicts hypotension during anesthesia induction. Acta Anaesthesiol Scand. 2010 May;54(5):596-602. doi: 10.1111/j.1399-6576.2010.02225.x. Epub 2010 Mar 10. PMID 20236098
- See also: The Effects of Motion on the Performance of Pulse Oximeters in Volunteers (Revised publication — https://doi.org/10.1097/00000542-199701000-00014